CLINICAL TRIAL: NCT05282537
Title: Evaluation of Mental Health, Sleep Quality, Level of Physical Activity, Food Intake, and Body Composition Before and After One Year of Face-to-face Academic Activities in University Students
Brief Title: Health Parameters of University Students After Pandemic Isolation
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Marco Antonio Hernández Lepe, Doctor, Universidad Autonoma de Baja California
Other Study IDs: UABC2022
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Mental Health Wellness 1; Sedentary Behavior
Keywords: Anxiety; Depression; Body composition; Food intake
MeSH Terms: conditions — Sedentary Behavior; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In person academic activities group: University students of health sciences area returning to in person academic activities in Mexico.
  All university students will return to in person academic activities in March, 2022, for that reason a limitation is that it is no possible to have a control group (Nobody is going to continue in virtual academic activities).
  Interventions: Behavioral: In person academic activities

INTERVENTIONS:
Behavioral: In person academic activities — All participants will perform academic activities in person from March to December, 2022

SUMMARY:
The COVID-19 pandemic caused by the SARS-CoV-2 coronavirus represents threats to global health and economy. The high pathogenesis of SARS-CoV-2 extent that the Mexican government declared a national health emergency, agreeing to take extraordinary measures such as the suspension of non-essential work, including the suspension of academic activities at all levels, in order to minimize the dispersion and transmission of the virus and its consequences. Several previously reported quarantine evaluations have shown that psychological stress reactions can arise from the experience of physical and social isolation, so the current global threat of isolation has shaken the usual practices of the general population, including young people, and resulting in the modification of their academic, labor and social dynamics.

The usual behavior in this phenomenon establishes that greater social isolation is associated with less satisfaction with life, higher levels of depression and lower levels of psychological well-being or performance as well as changes in diet. Understanding the factors related to coping with COVID-19 is essential to issue guidance on health in the student population, for that, the present proposal intends to evaluate changes in health parameters derived from the resumption of academic activities in person for a year in university students of health sciences area.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus (SARS-CoV-2) caused an outbreak of pneumonia of unknown origin in late December 2019, causing coronavirus disease 19 (COVID-19). After its high contagion capacity, a couple of weeks later the World Health Organization declared COVID-19 an international public security emergency, and by March 2020 it was officially declared a pandemic.

The rapid increase in the number of cases of infection and deaths from COVID-19 forced national governments to take extreme control and prevention measures. In Mexico, the community health strategy was defined in the "National Day of Healthy Distance", where the main guidelines included avoiding inter-personal contagion through confinement, forcing the suspension of all non-essential activities, which included the suspension of academic activities at all levels.

Although the measures that were taken to mitigate the spread of the disease are obtaining favorable results with respect to the transmission of the virus, but the modification of the academic, work, food and social dynamics are having an unprecedented impact on biological, psychological and social health of the population. In this sense, maintaining and promoting the physical and mental health of the population is a challenge that transcends the individual level and demands actions at the local, national and global levels.

Social isolation is a multidimensional event that contemplates both the quantity, as well as the inadequate quality of interactions with other people, including those not only in the family environment, but also at the community level. Social isolation has been studied mainly in older adults derived from their retirement or low mobility, however, the current global threat of isolation has shaken the usual practices of the general population, including young people and resulting in the modification of their academic, labor and social dynamics.

The usual behavior in this phenomenon establishes that greater social isolation is associated with lower life satisfaction, higher levels of depression and lower levels of psychological well-being or performance as well as changes in diet. The invitation to social isolation contemplated in the strategy of the Mexican government promoted the decrease in the level of physical activity in individuals during the last two years, while eating patterns were substantially modified by emotional and economic phenomena associated with each person. These levels of physical activity associated with food choices (voluntary or conditioned) have been shown to negatively affect health.

The lifestyle of university students prior to isolation due to the pandemic was already considered a risk factor for developing chronic non-communicable diseases, due to poor dietary intake, a low level of physical activity and a high level of sedentary lifestyle. Isolation has been shown to decrease physical activity levels and develop poor eating habits in North American university students, specifically in a study that included 125 participants, of which only 16% met the Canadian criteria for physical activity a week before of the pandemic, only 9.6% continued to comply with them during isolation. Furthermore, of the participants who did not meet the physical activity requirements, 55% showed a significant decrease in physical activity levels.

In response to the confinement due to the pandemic, clinically significant results have been reported regarding the presence of mental health problems such as acute stress and anguish in university students of health sciences area. This phenomenon has been attributed to the fact that students of health sciences area have a greater knowledge of COVID-19 (according to the general population), the risks associated with contracting it, symptoms and its possible social impact, for which may be more susceptible to develop mental health problems during the period of confinement.

In addition to confinement and physical inactivity, instability in the national economy contributes substantially to the genesis of mental health effects, such as fear, stress, and anxiety. The interplay between emotions and eating (referred to as emotional eating) has been addressed before, with evidence that changes in food intake are consistently the primary response during altered mental states.

ELIGIBILITY:
Inclusion Criteria:

* Health Sciences Students
* Informed consent sign

Exclusion Criteria:

* Fail a course by absences
* No assistance to evaluations

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 325 undergraduate students form the Medical and Phsychology School of the Autonomous University of Baja California will be invited to participate voluntarily.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Depression | March-December, 2022
  Patient Health Questionnaire (PHQ-7)
Physical activity | March-December, 2022
  International Physical Activity Questionnaire (IPAQ, short form)
Body fat percentage | March-December, 2022
  Air Displacement Plethysmography

SECONDARY OUTCOMES:
Anxiety | March-December, 2022
  General Anxiety Disorder 7 Questionnaire (GAD-7)
Sleep Quality | March-December, 2022
  Pittsburgh Sleep Quality Index (PSQI)
Body Mass Index | March-December, 2022
  Body Weight and Body Mass Evaluation
Waist to hip ratio | March-December, 2022
  Waist and hip girths
Food intake | March-December, 2022
  24 hour recalls

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Hernández-Lepe, Dr., Principal Investigator — Autonomous University of Baja California
Locations (1):
- Medical and Psychology School, Tijuana, California, Mexico

REFERENCES:
- [Background] World Health Organization. (2020). Mental health and psychosocial considerations during the COVID-19 outbreak, 18 March 2020 (No. WHO/2019-nCoV/MentalHealth/2020.1.
- [Background] Diario Oficial de la Federación, 2020. Acuerdo por el que se establecen las medidas preventivas que se deberán implementar para la mitigación y control de los riesgos para la salud que implica la enfermedad por el virus SARS-CoV2 (COVID-19). Visitado el 24 de febrero del 2022 en: https://www.dof.gob.mx/nota_detalle.php?codigo=5590339&fecha=24/03/2020.
- [Background] Prowse R, Sherratt F, Abizaid A, Gabrys RL, Hellemans KGC, Patterson ZR, McQuaid RJ. Coping With the COVID-19 Pandemic: Examining Gender Differences in Stress and Mental Health Among University Students. Front Psychiatry. 2021 Apr 7;12:650759. doi: 10.3389/fpsyt.2021.650759. eCollection 2021. PMID 33897499
- [Background] Gruber J, Prinstein MJ, Clark LA, Rottenberg J, Abramowitz JS, Albano AM, Aldao A, Borelli JL, Chung T, Davila J, Forbes EE, Gee DG, Hall GCN, Hallion LS, Hinshaw SP, Hofmann SG, Hollon SD, Joormann J, Kazdin AE, Klein DN, La Greca AM, Levenson RW, MacDonald AW, McKay D, McLaughlin KA, Mendle J, Miller AB, Neblett EW, Nock M, Olatunji BO, Persons JB, Rozek DC, Schleider JL, Slavich GM, Teachman BA, Vine V, Weinstock LM. Mental health and clinical psychological science in the time of COVID-19: Challenges, opportunities, and a call to action. Am Psychol. 2021 Apr;76(3):409-426. doi: 10.1037/amp0000707. Epub 2020 Aug 10. PMID 32772538
- [Background] Clair, R., Gordon, M., Kroon, M., & Reilly, C. (2021). The effects of social isolation on well-being and life satisfaction during pandemic. Humanities and Social Sciences Communications, 8(1), 1-6.
- [Background] Liu H, Zhang M, Yang Q, Yu B. Gender differences in the influence of social isolation and loneliness on depressive symptoms in college students: a longitudinal study. Soc Psychiatry Psychiatr Epidemiol. 2020 Feb;55(2):251-257. doi: 10.1007/s00127-019-01726-6. Epub 2019 May 21. PMID 31115597
- [Background] Dos Santos Quaresma MV, Marques CG, Magalhaes ACO, Dos Santos RVT. Emotional eating, binge eating, physical inactivity, and vespertine chronotype are negative predictors of dietary practices during COVID-19 social isolation: A cross-sectional study. Nutrition. 2021 Oct;90:111223. doi: 10.1016/j.nut.2021.111223. Epub 2021 Mar 9. PMID 33934054
- [Background] Martinez-Vazquez SE, Ceballos-Rasgado M, Posada-Velazquez R, Hunot-Alexander C, Nava-Gonzalez EJ, Ramirez-Silva I, Aguilar-Lopez DK, Quiroz-Olguin G, Lopez-Jara B, Delgado-de-la-Cruz C, Huescas-Juarez S, Silva M, Kaufer-Horwitz M. Perceived Diet Quality, Eating Behaviour, and Lifestyle Changes in a Mexican Population with Internet Access during Confinement for the COVID-19 Pandemic: ESCAN-COVID19Mx Survey. Nutrients. 2021 Nov 26;13(12):4256. doi: 10.3390/nu13124256. PMID 34959806
- [Background] Bertrand L, Shaw KA, Ko J, Deprez D, Chilibeck PD, Zello GA. The impact of the coronavirus disease 2019 (COVID-19) pandemic on university students' dietary intake, physical activity, and sedentary behaviour. Appl Physiol Nutr Metab. 2021 Mar;46(3):265-272. doi: 10.1139/apnm-2020-0990. Epub 2021 Jan 15. PMID 33449864
- [Background] Li Y, Wang Y, Jiang J, Valdimarsdottir UA, Fall K, Fang F, Song H, Lu D, Zhang W. Psychological distress among health professional students during the COVID-19 outbreak. Psychol Med. 2021 Aug;51(11):1952-1954. doi: 10.1017/S0033291720001555. Epub 2020 May 11. PMID 32389148
- [Background] Liu J, Zhu Q, Fan W, Makamure J, Zheng C, Wang J. Online Mental Health Survey in a Medical College in China During the COVID-19 Outbreak. Front Psychiatry. 2020 May 13;11:459. doi: 10.3389/fpsyt.2020.00459. eCollection 2020. PMID 32574242
- [Background] Reichenberger J, Kuppens P, Liedlgruber M, Wilhelm FH, Tiefengrabner M, Ginzinger S, Blechert J. No haste, more taste: An EMA study of the effects of stress, negative and positive emotions on eating behavior. Biol Psychol. 2018 Jan;131:54-62. doi: 10.1016/j.biopsycho.2016.09.002. Epub 2016 Sep 18. PMID 27654506